CLINICAL TRIAL: NCT01182181
Title: A Single-Dose, Comparative Bioavailability Study of Two Formulations of Anastrozole 1 mg Tablets Under Fasting Conditions
Brief Title: Anastrozole 1 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2005-1042
Record Dates: First submitted 2010-08-12; First posted 2010-08-16 (Estimated); Results first posted 2010-11-15 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-10

CONDITIONS: Healthy
Keywords: Healthy Subjects; Bioequivalence
MeSH Terms: interventions — Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational Test Product (Experimental): Anastrozole Tablets, 1 mg
  Interventions: Drug: Anastrozole (Teva Pharmaceuticals USA)
- Reference Listed Drug (Active Comparator): Arimidex® Tablets, 1 mg
  Interventions: Drug: Anastrozole (Arimidex®)

INTERVENTIONS:
Drug: Anastrozole (Teva Pharmaceuticals USA) — 1 mg Tablets
  Arms: Investigational Test Product
Drug: Anastrozole (Arimidex®) — 1 mg Tablets
  Other Names: Arimidex®
  Arms: Reference Listed Drug

SUMMARY:
The objective of this study is to evaluate the comparative bioavailability between Anastrozole 1 mg Tablets (Teva Pharmaceuticals USA) and Arimidex® 1 mg Tablets (AstraZeneca Pharmaceuticals LP, USA), after a single-dose in healthy subjects under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA Bioequivalence Statistical Methods

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking, post-menopausal or surgically sterile female subjects 18 years or age or older.
* Body mass index (BMI) between 19 and 30, inclusive.
* Indicate non-child bearing status by one of the following criteria:

  * Indication of successful hysterectomy.
  * No spontaneous menses for at least 1 year, must have luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels within postmenopausal range.
  * Indication of successful bilateral oophorectomy.
* Negative for:

  * HIV.
  * Hepatitis B surface antigen and Hepatitis C antibody.
  * Urine drugs of abuse test (marijuana, amphetamines, barbiturates, cocaine, opiates, benzodiazepines, and methadone).
  * Urine cotinine test.
  * Serum pregnancy test.
* No significant diseases or clinically significant findings in a physical examination.
* No clinically significant abnormal laboratory values.
* No clinically significant findings in the 12-lead electrocardiogram (ECG).
* No clinically significant findings from the vital signs measurement.
* Be informed of the nature of the study and given written consent prior to receiving any study procedure.
* Participants in this study will be unable to have children (i.e. post-menopausal, hysterectomy).

Exclusion Criteria:

* Known history or presence of any clinically significant medical condition.
* Known or suspected carcinoma.
* Known history of:

  * Hypersensitivity or idiosyncratic reaction to anastrozole and/or any other drug substances with similar activity.
  * Alcoholism within the last 12 months.
  * Drug dependence and/or substance abuse.
  * Use of tobacco or nicotine-containing products within the last 6 months.
* Taken any drug known to induce or inhibit hepatic drug metabolism in the 30 days prior to dosing.
* Taken any hormone replacement therapy (HRT) for 4 weeks prior to dosing.
* On a special diet within 4 weeks prior to drug administration (e.g. liquid, protein, raw food diet).
* Participated in another clinical trial or received an investigational product within 30 days prior to drug administration.
* Donated up to 250 mL of blood within the previous 30 days OR donated from 251 to 500 mL of blood in the previous 45 days OR donated more than 500 mL of blood in the previous 56 days.
* Requirement of any non-topical medication (prescription and/or over-the-counter) on a routine basis.
* Difficulty fasting or consuming the standard meals.
* Do not tolerate venipuncture.
* Unable to read or sign the informed consent form.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-08; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xueyu (Eric) Chen, M.D., Ph.D., FRCP, Principal Investigator — Pharma Medica Research, Inc.
Locations (1):
- Pharma Medica Research Inc., Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Anastrazole (Test) First: 1 mg Anastrozole Tablets test product dosed in first period followed by 1 mg Arimidex® Tablets reference product dosed in the second period.
- Arimidex® (Reference) First: 1 mg Arimidex® Tablets reference product dosed in first period followed by 1 mg Anastrazole Tablets test product dosed in the second period.
Period: First Intervention
Arm/Group | Anastrazole (Test) First | Arimidex® (Reference) First
Started | 11 | 11
Completed | 10 | 11
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout of 21 Days
Arm/Group | Anastrazole (Test) First | Arimidex® (Reference) First
Started | 10 | 11
Completed | 10 | 10
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention
Arm/Group | Anastrazole (Test) First | Arimidex® (Reference) First
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anastrazole (Test) First | Arimidex® (Reference) First | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 10 | 11 | 21
  Black | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Anastrozole(Maximum Observed Concentration of Drug Substance in Plasma)
Description: Bioequivalence based on Anastrozole Cmax.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Anastrazole (Test): 1 mg Anastrozole Tablets test product dosed in either period.
- Arimidex® (Reference): 1 mg Arimidex® Tablets reference product dosed in either period.
Arm/Group | Anastrazole (Test) | Arimidex® (Reference)
Number analyzed (Participants) | 20 | 20
ng/mL | 17.1 (3.3) | 17.8 (2.7)
Statistical Analysis 1: Comparison: Anastrazole (Test) vs Arimidex® (Reference); Test type: Non-Inferiority or Equivalence — ANOVA is to be used to identify the source contributions by factors including subjects, period, formulation and potential interactions. The geometric mean ratio together with the ANOVA residual mean error term are used to identify the statistical basis for the 90% confidence interval for the ratio of the population means (Test [T]/Reference[R]) of the identified metrics (e.g. AUC, Cmax); Ratio of the T/R geometric mean x 100 = 95.6, 90% CI 2-sided [92.34 to 98.95] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference (R) and test (T) product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t of Anastrozole(Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on Anastrozole AUC0-t.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Anastrazole (Test) | Arimidex® (Reference)
Number analyzed (Participants) | 20 | 20
ng*h/mL | 503 (110) | 519 (94)
Statistical Analysis 1: Comparison: Anastrazole (Test) vs Arimidex® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 96.3, 90% CI 2-sided [93.14 to 99.57] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study, which was approximately 6 weeks in duration.
Description: Volunteers were monitored throughout the study for any adverse experiences. AEs were collected through both solicited and unsolicited methods. The volunteers were encouraged to report signs, symptoms, and any changes in health to the clinic staff.
Arm/Group | Anastrazole (Test) | Arimidex® (Reference)
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 2/22 | 4/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anastrazole (Test) (N=22) | Arimidex® (Reference) (N=22)
Hematuria (General disorders) | 2 (4) | 1 (2)
Abnormal Urine (General disorders) | 2 (5) | 1 (3)
Headache (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.